CLINICAL TRIAL: NCT06961136
Title: Prospective Cohort Study on Fuzheng Yangxin Prescription For Rapid Rehabilitation of Patients With Qi-Yin Deficiency Syndrome After Coronary Artery Bypass Grafting
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BYSY202451303
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Bypass
Keywords: Coronary Artery Bypass; Chinese herbal medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fuzheng Yangxin prescription
  Interventions: Drug: Fuzheng Yangxin prescription
- placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Fuzheng Yangxin prescription — Fuzheng Yangxin prescription
  Groups: Fuzheng Yangxin prescription
Drug: placebo — placebo
  Groups: placebo

SUMMARY:
Data from the Global Burden of Disease Study 2021, recently published in the Lancet, show that ischaemic heart disease remains the first most common cause of death worldwide. Ischemic heart disease mainly refers to coronary artery stenosis or obstruction caused by coronary artery atherosclerosis leading to myocardial ischemia heart disease, called coronary heart disease. "China Cardiovascular Health and Disease Report 2022" mentioned that coronary heart disease is an important cardiovascular disease affecting the health of Chinese residents, and its prevalence and mortality are on the rise. Coronary artery bypass grafting (CABG) and interventional therapy (PCI) are commonly used in the treatment of coronary heart disease. CABG surgery can significantly reduce the recurrence of angina pectoris, the incidence of acute myocardial infarction and improve the survival rate of patients, the patency rate of 5 years after mammary arterial bridge can reach more than 90%. Current guidelines and various RCT studies have shown that CABG is the gold standard for revascularization in patients with complex coronary artery disease. With the increasing aging of Chinese population, there are more and more cases of complex coronary artery diseases, and CABG, as the first choice for complex coronary artery diseases, will be more and more widely used in the foreseeable future. At present, the number of coronary artery bypass surgery is on the rise, about 50,000 cases per year. Traditional Chinese medicine can play a role in preventing complications, improving the quality of life and long-term curative effect of patients after CABG. It is particularly important to actively seek the treatment of integrated Chinese and Western medicine for patients after CABG. This study aims to explore the effectiveness and safety of Fuzheng Yangxin prescription in the treatment of Qi-Yin deficiency after CABG by means of a prospective cohort study, so as to determine the efficacy of Fuzheng Yangxin prescription on the recovery after CABG. To formulate a routine program of Chinese and Western combined therapy for postoperative rehabilitation of cardiac surgery, and actively promote the technology and program, promote the transformation of intellectual property rights, etc., and contribute to the formulation of relevant guidelines.

DETAILED DESCRIPTION:
Data from the Global Burden of Disease Study 2021, recently published in the Lancet, show that ischaemic heart disease remains the first most common cause of death worldwide. Ischemic heart disease mainly refers to coronary artery stenosis or obstruction caused by coronary artery atherosclerosis leading to myocardial ischemia heart disease, called coronary heart disease. "China Cardiovascular Health and Disease Report 2022" mentioned that coronary heart disease is an important cardiovascular disease affecting the health of Chinese residents, and its prevalence and mortality are on the rise. Coronary artery bypass grafting (CABG) and interventional therapy (PCI) are commonly used in the treatment of coronary heart disease. CABG surgery can significantly reduce the recurrence of angina pectoris, the incidence of acute myocardial infarction and improve the survival rate of patients, the patency rate of 5 years after mammary arterial bridge can reach more than 90%. Current guidelines and various RCT studies have shown that CABG is the gold standard for revascularization in patients with complex coronary artery disease. With the increasing aging of Chinese population, there are more and more cases of complex coronary artery diseases, and CABG, as the first choice for complex coronary artery diseases, will be more and more widely used in the foreseeable future. At present, the number of coronary artery bypass surgery is on the rise, about 50,000 cases per year.

Although CABG surgery has a better long-term survival rate for patients with complex lesions, no matter what method of CABG surgery, it will inevitably cause a large blow to patients and bring a huge burden on patients' physiological and psychological functions in the early postoperative period. In the SYNTAX trial, The physiological function scores (SF-36 and EQ-5D) of the patients after CABG were significantly lower than those after PCI. Another RCT study, the FREEDOM trial, showed that although CABG had a good quality of life and physiological status 12 months after surgery, compared with PCI, CABG quality of life and psychological status scores were significantly lower at 6 months after surgery. These trials suggest that patients with CABG face an early recovery challenge due to surgical trauma. And as the number of older adults receiving CABG increases, the problem is likely to get worse. At the same time, there are many postoperative complications such as myocardial infarction, heart failure and atrial fibrillation after CABG.

Traditional Chinese medicine can play a role in preventing complications, improving the quality of life and long-term curative effect of patients after CABG. It is particularly important to actively seek the treatment of integrated Chinese and Western medicine for patients after CABG. This study aims to explore the effectiveness and safety of Fuzheng Yangxin prescription in the treatment of Qi-Yin deficiency after CABG by means of a prospective cohort study, so as to determine the efficacy of Fuzheng Yangxin prescription on the recovery after CABG. To formulate a routine program of Chinese and Western combined therapy for postoperative rehabilitation of cardiac surgery, and actively promote the technology and program, promote the transformation of intellectual property rights, etc., and contribute to the formulation of relevant guidelines.

If this study confirms the effectiveness and safety of Fuzheng Yangxin prescription in treating Qi-Yin deficiency syndrome after CABG operation, it can significantly improve patients' quality of life and shorten hospitalization and rehabilitation time, which can benefit more patients, significantly reduce medical costs and reduce the burden of medical insurance, and contribute to the implementation of the Healthy China strategy. At the same time, through the promotion of this project, it is expected to promote the cooperation between traditional Chinese and Western medicine after cardiac surgery, form a routine program and promote it, accelerate the transformation of intellectual property rights, and promote the construction of the "flagship" hospital of traditional Chinese and Western medicine cooperation in Peking University Third Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received coronary artery bypass surgery with syndrome differentiation of Qi-Yin deficiency after operation

Exclusion Criteria:

* ① Patients allergic to Fuzheng Yangxin Fang granules

  * Patients with postoperative cold and fever ③ Patients with severe postoperative hepatic and renal insufficiency ④ Other circumstances: Concurrent valvular surgery or other cardiac surgery, end-stage malignant tumor, uncontrolled infection, bleeding, progressive degenerative systemic disease, severe brain injury, multiple organ failure, other vital organ dysfunction such as severe liver impairment, severe heart failure or cardiogenic shock, inability to tolerate surgery, etc.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received coronary artery bypass surgery with syndrome differentiation of Qi-Yin deficiency after operation
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
SAQ scores on PL | 7days

SECONDARY OUTCOMES:
Perioperative safety index | 14d
SAQ scores on others | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No